CLINICAL TRIAL: NCT03106311
Title: Use of Beta Subunit of Human Chorionic Gonadotropin Assay as a Diagnostic Tool for Premature Rupture of Membranes
Brief Title: The Use of Quantitative Pregnancy Test in Amniotic Fluid as a Diagnostic Tool for Rupture of Fetal Membranes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Omran, Principal investigator, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 4567
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Premature Rupture of Membrane
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rupture of membranes group (Active Comparator): Pregnant women with definite rupture of membranes will undergo speculum examination. Vaginal washing will be done. The washing fluid will be taken for quantitative and qualitative assessment of beta subunit of human chorionic gonadotropin.
  Interventions: Diagnostic Test: assessment of beta subunit of human chorionic gonadotropin
- Intact membranes group (Active Comparator): Pregnant women with intact membranes will undergo speculum examination. Vaginal washing will be done. The washing fluid will be taken for quantitative and qualitative assessment of beta subunit of human chorionic gonadotropin.
  Interventions: Diagnostic Test: assessment of beta subunit of human chorionic gonadotropin

INTERVENTIONS:
Diagnostic Test: assessment of beta subunit of human chorionic gonadotropin — Vaginal washing fluid will be collected and sent for measurement of beta subunit of human chorionic gonadotropin

SUMMARY:
Two groups will be recruited. The first group are pregnant ladies that have unequivocal rupture of fetal membranes that is diagnosed by seeing the amniotic fluid leakage in the vagina. The second group are normal pregnant ladies without rupture of membranes. both groups will be tested by taking vaginal washing fluid. Quantitative and qualitative pregnancy tests will be measured in this fluid.

DETAILED DESCRIPTION:
Beta subunit of human chorionic gonadotropin assay will be measured in the vaginal washing in two groups. The first group are pregnant women in the second or third trimester. These women have definite rupture of membranes diagnosed by visual leaking of the amniotic fluid from the cervix during speculum examination. The second group are pregnant women with intact membranes. Assessment of both the qualitative and quantitative beta subunit of human chorionic gonadotropin will be done

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 14 and 40 weeks gestation with history of gush of vaginal fluid
* Pregnant women between without history of gush of vaginal fluid

Exclusion Criteria:

* Presence of vaginal bleeding
* Presence of any obstetric emergency as cord prolapse

Ages: 17 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Concentration of beta subunit of human chorionic gonadotropin | This outcome will be measured within 20 minutes of collection of vaginal washing fluid. The collection of vaginal washing fluid will be done by an investigator upon admission to the department of Obstetrics
  Concentration of beta subunit of human chorionic gonadotropin will be measured in vaginal washing fluid. The collection of vaginal washing fluid will be done by an investigator

SECONDARY OUTCOMES:
Presence or absence of positive qualitative pregnancy test | Qualitative pregnancy test will be done in the vaginal washing fluid by an investigator within 20 minutes from admission to the Obstetrics department.
  Qualitative pregnancy test will be done by an investigator in the Obstetrics department

CONTACTS AND LOCATIONS:
Overall Officials: Eman Omran, M.D., Principal Investigator — Cairo University
Locations (1):
- Department of Obstetrics and Gynecology, Kasr Al-Ainy hospital, Cairo, Greater Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided